CLINICAL TRIAL: NCT06019715
Title: Remote Postpartum Intervention Targeting Movement Behaviors After Hypertensive Disorders of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jackie Dziewior (Other)
Responsible Party: Sponsor-Investigator, Jackie Dziewior, PhD Candidate, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202302470
Record Dates: First submitted 2023-08-24; First posted 2023-08-31 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Hypertensive Disorder of Pregnancy
MeSH Terms: conditions — Toxemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): This arm will receive the full intervention, including 4 months of health coaching support, 8 virtual health coaching visits, a Fitbit device, and an at home blood pressure monitor.
  Interventions: Behavioral: Postpartum Remote Physical Activity Intervention

INTERVENTIONS:
Behavioral: Postpartum Remote Physical Activity Intervention — Includes 8 remote health coaching session to promote physical activity, use of a Fitbit device, and use of a home based blood pressure monitor.
  Other Names: The HyPE Intervention

SUMMARY:
The purpose of this study is to test the feasibility, acceptability, and preliminary efficacy of a postpartum physical activity intervention after a pregnancy complicated by a Hypertensive Disorder of Pregnancy. The study will also assess the effects of the remote postpartum intervention on blood pressure. To do this, we will recruit individuals that are 3-6 months postpartum a pregnancy complicated by a hypertensive disorder to participate in a 4-month health coaching intervention aimed to promote physical activity and was informed by formative work done previously.

DETAILED DESCRIPTION:
I.a Clinical and Public Health Significance. CVD is the leading cause of death among women in America; one in four of these deaths are preventable.3 HDP, including gestational and chronic hypertension, preeclampsia, and superimposed preeclampsia, are risk factors for CVD.3 HDP are associated with maternal and offspring morbidity and mortality, negatively impacting cardiovascular, immune, and neurological systems.21 With 10% of all pregnancies affected by HDP, targeting this population is critical to improving maternal/neonatal morbidity and mortality and overall cardiovascular health in America.1,2 The proposed study answers the AHA's call in their 2022 scientific statement for studies demonstrating efficacy of lifestyle interventions addressing hypertension during the postpartum period among those with HDP.22

I.b Cardiovascular changes during pregnancy act as a natural stress test and may uncover an individual's potential risk of future CVD.23 Specifically, individuals with HDP are at an immediately increased risk for HTN after delivery.1 Long-term cardiometabolic health is also implicated by HDP, with increased risk of future CVD, morbidity, and mortality compared to normotensive pregnancies.24 Odds of developing HTN at one year postpartum is 12 to 25 times greater in HDP pregnancies compared to normotensive pregnancies.25 The 5-year likelihood of developing HTN for pregnancies complicated by HDP is 7.1 times greater than normotensive pregnancies.1 Even in those not diagnosed with HTN, the BP is on average greater in HDP women than in normotensive pregnancies.26

I.c Follow-up care for HDP in the postpartum period is inadequate. Although it is understood that HDP place an individual at increased risk for future CVD, only 58% of women with HDP had a 7-10 day postpartum BP check and 48% for a 6-month postpartum visit.4,25 In addition, only 17% of women with HDP follow-up with their primary care providers, indicating a gap in the transition of care after pregnancy.25 Lack of follow-up has been attributed to fatigue, pain, infant care obligations, time, and low awareness of HDP as a risk factor for future CVD.27,28 Although a few interventions have targeted future CVD risk in this population, few to no studies account for these unique barriers experienced during the postpartum period.14,29

I.d PA and SED have independent effects on CVD risk.8-10 PA and SED are modifiable risk factors for CVD and have the potential to improve BP.30 Current studies suggest that moderate to vigorous PA decreases after pregnancy, and evidence concerning SED is conflicting.31,32 PA, specifically aerobic exercise, has beneficial effects on mean, systolic, and diastolic BP in adults.33,34 This association has been observed in pregnant populations as well, with the greatest improvements seen in inactive individuals.35,36 SED is another modifiable risk factor associated with CVD, independent of PA, with each additional hour of SED increasing the risk for HTN.8 Although the effect on PA and SED in the general population are well understood, the direct effects of PA/SED in the postpartum period on BP after HDP is understudied.37

I.e The perinatal period presents a critical period of change and a promising target for lifestyle intervention to reduce future CVD risk. The association of HDP with future CVD elicited AHA's call to action for more vigorous primary prevention of CVD in the postpartum period.38,39 With increased contact to health care professionals during gestation, pregnancy also offers an opportunity to connect with this population to develop positive health behaviors, which our preliminary data confirms is feasible. Interventions promoting PA and decreased SED in the postpartum period after a HDP is an under explored primary prevention strategy.37

ELIGIBILITY:
Inclusion Criteria:

* <6 months postpartum from a pregnancy complicated by a hypertensive disorder
* Have self-reported insufficient activity (<150 minutes of moderate to vigorous physical activity per week)
* Own a smartphone

Exclusion Criteria:

* Current enrollment in another physical activity or sedentary behavior intervention study
* Recommend to limit physical activity by a healthcare provider
* Diagnosed with diabetes, kidney disease, cardiovascular disease
* Prior bariatric surgery
* Currently takes medication to reduce weight or anti-hypertensives

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Change in physical activity | 6 months
  Change in step count from baseline across study timeline
Intervention feasibility | 6 months
  Will be evaluated using Bowen's standards, specifically implementation and practicality. Implementation and practicability will be measured by the number of completed sessions out of the total session possible and by the quality of implementation through participant self-reported satisfaction of the program's session length, frequency, and topics covered.
Intervention acceptability | 6 months
  Will be evaluated using Bowen's standards, specifically acceptability and demand of the intervention. Acceptability and demand will be assessed by participant self-reported satisfaction and likelihood to recommend the program to other of participants. Acceptability, demand, and practicality will be defined by at least 75% of participants responding either satisfied or very satisfied to these questions; implementation by 75% of sessions attended.

SECONDARY OUTCOMES:
Change in postpartum blood pressure | 6 months
  Change in postpartum blood pressure from baseline across study timeline

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melchiorre K, Thilaganathan B, Giorgione V, Ridder A, Memmo A, Khalil A. Hypertensive Disorders of Pregnancy and Future Cardiovascular Health. Front Cardiovasc Med. 2020 Apr 15;7:59. doi: 10.3389/fcvm.2020.00059. eCollection 2020. PMID 32351977
- [Background] Diaz KM, Shimbo D. Physical activity and the prevention of hypertension. Curr Hypertens Rep. 2013 Dec;15(6):659-68. doi: 10.1007/s11906-013-0386-8. PMID 24052212
- [Background] Evenson KR, Aytur SA, Borodulin K. Physical activity beliefs, barriers, and enablers among postpartum women. J Womens Health (Larchmt). 2009 Dec;18(12):1925-34. doi: 10.1089/jwh.2008.1309. PMID 20044854
- [Background] Lane-Cordova AD, Jerome GJ, Paluch AE, Bustamante EE, LaMonte MJ, Pate RR, Weaver RG, Webber-Ritchey KJ, Gibbs BB; Committee on Physical Activity of the American Heart Association Council on Lifestyle and Cardiometabolic Health. Supporting Physical Activity in Patients and Populations During Life Events and Transitions: A Scientific Statement From the American Heart Association. Circulation. 2022 Jan 25;145(4):e117-e128. doi: 10.1161/CIR.0000000000001035. Epub 2021 Dec 1. PMID 34847691
- [Background] Lui NA, Jeyaram G, Henry A. Postpartum Interventions to Reduce Long-Term Cardiovascular Disease Risk in Women After Hypertensive Disorders of Pregnancy: A Systematic Review. Front Cardiovasc Med. 2019 Nov 15;6:160. doi: 10.3389/fcvm.2019.00160. eCollection 2019. PMID 31803757
- [Background] Whitaker KM, Jones MA, Dziewior J, Anderson M, Anderson C, Gibbs BB, Carr LJ. Feasibility, acceptability, and preliminary efficacy of a single-arm, remotely-delivered health coaching intervention to increase physical activity and reduce sedentary behavior during pregnancy. BMC Pregnancy Childbirth. 2022 Oct 2;22(1):740. doi: 10.1186/s12884-022-05073-4. PMID 36184599
- [Background] Whelton SP, Chin A, Xin X, He J. Effect of aerobic exercise on blood pressure: a meta-analysis of randomized, controlled trials. Ann Intern Med. 2002 Apr 2;136(7):493-503. doi: 10.7326/0003-4819-136-7-200204020-00006. PMID 11926784
- [Background] Hutchesson M, Campbell L, Leonard A, Vincze L, Shrewsbury V, Collins C, Taylor R. Do modifiable risk factors for cardiovascular disease post-pregnancy influence the association between hypertensive disorders of pregnancy and cardiovascular health outcomes? A systematic review of observational studies. Pregnancy Hypertens. 2022 Mar;27:138-147. doi: 10.1016/j.preghy.2021.12.017. Epub 2022 Jan 6. PMID 35066405
- [Background] Mehta LS, Sharma G, Creanga AA, Hameed AB, Hollier LM, Johnson JC, Leffert L, McCullough LD, Mujahid MS, Watson K, White CJ; American Heart Association Advocacy Coordinating Committee. Call to Action: Maternal Health and Saving Mothers: A Policy Statement From the American Heart Association. Circulation. 2021 Oct 12;144(15):e251-e269. doi: 10.1161/CIR.0000000000001000. Epub 2021 Sep 8. PMID 34493059